CLINICAL TRIAL: NCT03513133
Title: Rehabilitation of Working Memory After Traumatic Brain Injury: Pilot Study of Brain Plasticity in Multimodal Advanced MRI
Brief Title: Rehabilitation of Working Memory and Brain Plasticity After Traumatic Brain Injury: Plastim-MDTC
Acronym: Plastim-MDTC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A00678-43
Record Dates: First submitted 2018-02-19; First posted 2018-05-01 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-02

CONDITIONS: Traumatic Brain Injury; Cognitive Impairment
Keywords: working memory; cognitive rehabilitation; functional neuroimaging
MeSH Terms: conditions — Brain Injuries, Traumatic; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: a group of 10 patients with severe TBI will receive 3-month rehabilitation of working memory and will be compared to a group of 10 healthy controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- working memory training (Experimental): Patients with severe TBI will receive a hierarchical training of working memory according to a previously described methodology. They will receive 3 sessions per week during three months (each session=1 h approximately)
  Interventions: Behavioral: working memory training

INTERVENTIONS:
Behavioral: working memory training — Hierarchical cognitive training of the different components of working memory according to Baddeley model; 15 tasks are used addressing: the phonological loop (8 tasks), the visuospatial sketchpad (4 tasks) and the central executive 3 tasks). Task are given in a hierarchical order, according to each individual patient's deficits and improvement.

SUMMARY:
The aim of this study is to assess the brain correlates, as assessed with multimodal MRI, of working memory training in patients with severe traumatic brain injury (TBI)

DETAILED DESCRIPTION:
This is a pilot feasibility study. Patients with subacute/chronic (> 6 months) severe TBI will be included if they suffer from a deficit in working memory. They will receive a specific hierarchical training of working memory (3 sessions per week during three months), according to a previously described methodology.

A multimodal MRI will be performed at neuroSpin center (CEA, Orsay, France) before and after cognitive training, including: structural imaging (T1, FLAIR and diffusion tensor imaging, DTI); functional connectivity at rest; and functional activation during a working memory task (n-back).

Behavioral and imaging changes after training will be analysed individually and compared to a group of healthy controls matched for age, gender and education.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe traumatic brain injury
* 6 months or more after the injury
* working memory deficit on cognitive testing

Exclusion Criteria:

* previous neurological or psychiatric condition
* severe behavioral troubles
* contra-indication to MRI
* pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
working memory questionnaire | change from baseline to 3 months
  It is a self-assessment questionnaire comprising 30 questions scored on a five-point Likert scale, ranging from 0 ("no problem at all") to 4 ("very severe problem in everyday life"). The total score will be used.

SECONDARY OUTCOMES:
working memory testing | change from baseline to 3 months
  neuropsychological assessment of working memory
neuro-imaging changes | change from baseline to 3 months
  multimodal 3T MRI

CONTACTS AND LOCATIONS:
Overall Officials: Philippe AZOUVI, MD-PhD, Study Chair — APHP Hôpital Raymond Poincaré; Lucie HERTZ PANNIER, MD, Principal Investigator — Neurospin- CEA; Eric BRUNET, MD, Principal Investigator — Hôpital André Mignot; Claire Vallat-Azouvi, PhD, Principal Investigator — University of Paris 8
Locations (1):
- APHP Hôpital Raymond Poincaré, Garches, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vallat C, Azouvi P, Hardisson H, Meffert R, Tessier C, Pradat-Diehl P. Rehabilitation of verbal working memory after left hemisphere stroke. Brain Inj. 2005 Dec;19(13):1157-64. doi: 10.1080/02699050500110595. PMID 16286329
- [Background] Vallat-Azouvi C, Pradat-Diehl P, Azouvi P. The Working Memory Questionnaire: a scale to assess everyday life problems related to deficits of working memory in brain injured patients. Neuropsychol Rehabil. 2012;22(4):634-49. doi: 10.1080/09602011.2012.681110. Epub 2012 Apr 27. PMID 22537095
- [Background] Vallat-Azouvi C, Pradat-Diehl P, Azouvi P. Rehabilitation of the central executive of working memory after severe traumatic brain injury: two single-case studies. Brain Inj. 2009 Jun;23(6):585-94. doi: 10.1080/02699050902970711. PMID 19484632
- [Background] Vallat-Azouvi C, Pradat-Diehl P, Azouvi P. Modularity in rehabilitation of working memory: a single-case study. Neuropsychol Rehabil. 2014;24(2):220-37. doi: 10.1080/09602011.2014.881294. Epub 2014 Feb 19. PMID 24552571